CLINICAL TRIAL: NCT02300636
Title: Randomized-controlled,Resistive Co-contraction Training Enhances Strength Recovery After Anterior Cruciate Ligament Reconstruction
Brief Title: Resistive Co-contraction Training After Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, GULCAN HARPUT, PT, MSc, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 014T03102002
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Muscle Weakness
Keywords: Knee joint; Muscle strength; anterior cruciate ligament
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Training: open kinetic (Experimental): Co-contraction training in open kinetic chain position
  8 weeks, 3 days in a week
  Interventions: Other: Training
- Training: closed kinetic (Experimental): Co-contraction training in closed kinetic chain position
  8 weeks, 3 days in a week
  Interventions: Other: Training
- Training: Standard ACL rehabilitation (Active Comparator): Standard ACL rehabilitation
  8 weeks, 3 days in a week
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — Co-contraction training at 60 knee flexion angle by using isokinetic dynamometer
  Arms: Training: open kinetic
Other: Training — Co-contraction training at 60 knee flexion angle by using leg press machine
  Arms: Training: closed kinetic
Other: Training — Standard ACL rehabilitation
  Arms: Training: Standard ACL rehabilitation

SUMMARY:
This study investigates different resistive co-contraction trainings effect on knee strength recovery after ACL reconstruction. Participants will be divided into three groups. Group 1 will receive standard ACL rehabilitation with 8 week co-contraction training in open kinetic chain position, Group 2 will receive standard ACL rehabilitation with 8 week co-contraction training in open kinetic chain position and Group 3 (control group) will only receive standard ACL rehabilitation.

DETAILED DESCRIPTION:
Co-contraction trainings can enhance joint stability via improving proprioceptive ability and stimulates muscle activity after injury and/or surgery. The participants will be assigned to the different groups one month after surgery. They will receive 8-week-treatment. Isometric strength of quadriceps and hamstring muscles will be measured at first,third and sixth months after surgery. Concentric and eccentric strength of quadriceps and hamstring muscles will be measured only at sixth months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ACL reconstruction with hamstring autograft
* starting PT program within one week after surgery

Exclusion Criteria:

* Revision surgery
* serious cartilage damage and/or cartilage repair
* ACL reconstruction with allograft and patellar tendon graft
* Having systemic and/or neurological problems

Ages: 17 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
knee muscle strength recovery | 8 weeks
  isometric, concentric and eccentric strength

SECONDARY OUTCOMES:
hamstring quadriceps ratio | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GULCAN HARPUT, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Cho SH, Bae CH, Gak HB. Effects of closed kinetic chain exercises on proprioception and functional scores of the knee after anterior cruciate ligament reconstruction. J Phys Ther Sci. 2013 Oct;25(10):1239-41. doi: 10.1589/jpts.25.1239. Epub 2013 Nov 20. PMID 24259766
- [Background] Lobb R, Tumilty S, Claydon LS. A review of systematic reviews on anterior cruciate ligament reconstruction rehabilitation. Phys Ther Sport. 2012 Nov;13(4):270-8. doi: 10.1016/j.ptsp.2012.05.001. Epub 2012 Jun 7. PMID 23068905
- [Background] Begalle RL, Distefano LJ, Blackburn T, Padua DA. Quadriceps and hamstrings coactivation during common therapeutic exercises. J Athl Train. 2012 Jul-Aug;47(4):396-405. doi: 10.4085/1062-6050-47.4.01. PMID 22889655
- [Background] Glass R, Waddell J, Hoogenboom B. The Effects of Open versus Closed Kinetic Chain Exercises on Patients with ACL Deficient or Reconstructed Knees: A Systematic Review. N Am J Sports Phys Ther. 2010 Jun;5(2):74-84. PMID 21589664
- [Background] Tagesson S, Oberg B, Good L, Kvist J. A comprehensive rehabilitation program with quadriceps strengthening in closed versus open kinetic chain exercise in patients with anterior cruciate ligament deficiency: a randomized clinical trial evaluating dynamic tibial translation and muscle function. Am J Sports Med. 2008 Feb;36(2):298-307. doi: 10.1177/0363546507307867. Epub 2007 Oct 16. PMID 17940146
- [Background] Biscarini A, Benvenuti P, Botti FM, Brunetti A, Brunetti O, Pettorossi VE. Voluntary enhanced cocontraction of hamstring muscles during open kinetic chain leg extension exercise: its potential unloading effect on the anterior cruciate ligament. Am J Sports Med. 2014 Sep;42(9):2103-12. doi: 10.1177/0363546514536137. Epub 2014 Jun 10. PMID 24918112
- [Background] Palmieri-Smith RM, McLean SG, Ashton-Miller JA, Wojtys EM. Association of quadriceps and hamstrings cocontraction patterns with knee joint loading. J Athl Train. 2009 May-Jun;44(3):256-63. doi: 10.4085/1062-6050-44.3.256. PMID 19478837